CLINICAL TRIAL: NCT02573220
Title: A UGT1A1 Genotype-Guided Dosing Study of Irinotecan Administered in Combination With 5-Fluorouracil/Leucovorin (FOLFIRI) and Cetuximab as First-Line Therapy in RAS Wild-Type Metastatic Colorectal Cancer Patients
Brief Title: Irinotecan Hydrochloride With FOLFIRI and Cetuximab as First-Line Therapy in Treating Patients With RAS Wild-Type Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated by PI due to inability to accrue.
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-0081; NCI-2015-01432 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB15-0081 (Other: University of Chicago Comprehensive Cancer Center); P30CA014599 (NIH)
Record Dates: First submitted 2015-09-21; First posted 2015-10-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (FOLFIRI and cetuximab) (Experimental): Patients receive irinotecan hydrochloride IV over 1-2 hours, fluorouracil IV continuously over 46 hours, and leucovorin calcium IV on days 1 and 15. Patients also receive cetuximab IV over 2 hours on days 3 and 15 of course 1 and days 1 and 15 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Erbitux
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluorouracil; 5-FU
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Camptosar; Camptothecin 11
Drug: Leucovorin Calcium — Given IV
  Other Names: Calcifolin; Wellcovorin

SUMMARY:
This phase I trial studies the side effects and the best dose of irinotecan hydrochloride, based on a genetic test, when given in combination with fluorouracil, leucovorin calcium, and cetuximab as first-line therapy in treating patients with an abnormal gene called RAS wild-type that has spread to other parts of the body (metastatic). Patients may also have a gene called uridine diphosphate glucuronosyltransferase (UGT1A1) that may interfere with the way irinotecan hydrochloride is absorbed by the body and may not be able to tolerate it. Determining the presence of this gene may help determine the best dose of irinotecan hydrochloride when given with fluorouracil and leucovorin calcium (FOLFIRI). Combination chemotherapy, such as FOLFIRI, works in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Cetuximab may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving FOLFIRI together with cetuximab may be a better treatment for patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD), the dose limiting toxicity (DLT) and the phase II recommended dosage of irinotecan (irinotecan hydrochloride) administered in the FOLFIRI regimen plus cetuximab in metastatic colorectal cancer (mCRC) patients with *1/*1 and *1/*28 uridine diphosphate glucuronosyltransferase (UGT1A1) genotype treated as first line chemotherapy.

SECONDARY OBJECTIVE:

To estimate the response rate, progression-free survival (PFS) and metastasectomy (with curative intent) rate in the overall patient population (both genotype cohorts).

OTHER OBJECTIVES:

I. To evaluate the variability of irinotecan pharmacokinetics, in combination with cetuximab, in patients with *1/*1 and *1/*28 genotype and the effect of the pharmacokinetic profile on toxicity and response rate.

II. To evaluate the pharmacokinetic profile of irinotecan and its major metabolites in the absence and the presence of cetuximab administration, in order to define the effect of the chimeric monoclonal antibody on irinotecan pharmacokinetics.

OUTLINE: This is a dose-escalation study of irinotecan hydrochloride in patients with UGT1A1.

Patients receive irinotecan hydrochloride intravenously (IV) over 1-2 hours, fluorouracil IV continuously over 46 hours, and leucovorin calcium IV on days 1 and 15. Patients also receive cetuximab IV over 2 hours on days 3 and 15 of course 1 and days 1 and 15 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of mCRC
* RAS wild-type status (by a Clinical Laboratory Improvement Amendments [CLIA] certified assay that includes all known mutations in Kirsten rat sarcoma viral oncogene homolog [KRAS], Harvey rat sarcoma viral oncogene homolog [HRAS], and neuroblastoma RAS viral (v-ras) oncogene homolog [NRAS])
* No prior chemotherapy for metastatic disease
* Able to understand and provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy > 3 months
* Measurable or evaluable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) criteria, i.e. lesions that can be accurately measured in at least one dimension with the longest diameter >= 20 mm using conventional techniques or >= 10 mm using spiral computed tomography (CT) scan
* Absolute neutrophil count (ANC) > l500/ul
* Hemoglobin > 9g/dL
* Platelets > 100,000/ul
* Total bilirubin =< 1.5 times upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal
* Alkaline phosphatase < 2.5 times the upper limit of normal, unless bone metastasis is present in the absence of liver metastasis
* Creatinine < 1.5 mg/dL
* Patients genotyped for UGT1A1*28 polymorphism with *1/*1 or *1/*28 genotype
* Men and women of childbearing potential must agree to use adequate contraception (double barrier birth control) for the duration of study therapy
* Negative serum or urine beta-human chorionic gonadotropin (hCG) pregnancy test at screening for patients of childbearing potential

Exclusion Criteria:

* Patients with both variant alleles (*28/*28)
* Patients with any polymorphism in UGT1A1 other than *1 or *28 (e.g, *6)
* Uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months prior to study treatment, New York Heart Association (NYHA) class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease or cardiac amyloidosis
* Patients with specific contraindications to the use of anti-EGFR therapy such as pulmonary fibrosis, interstitial pneumonia history
* Unresolved diarrhea and bowel obstruction
* Active bleeding
* Documented cerebral metastasis
* Serious active infectious disease
* Pregnancy
* Radiotherapy or major surgery within 4 weeks
* Psychiatric illness or social situations that would limit compliance with study requirements
* Presence of previous or concomitant neoplasm with exclusion of in situ cervical cancer
* Patients taking substrates, inhibitors and inducers of CYP3A4 should be encouraged to switch to alternative drugs whenever possible, given the potential for drug-drug interactions with irinotecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  The MTD recommended for phase II studies will be defined as the dose level immediately below the one at which 1 out of 3 patients or 1 out of 6 patients experienced DLT. Therefore at the MTD, 1/3 out of at least 10 patients experienced DLT. No intra-patient dose escalation is allowed. There will be two genotype cohorts of patients: one for each genotype. The cumulative hematological and non-hematological toxicities as well as the number of dose reductions and a delay in starting the next cycle of treatment will be used as secondary indicators to differentiate the two genotype cohorts of patients. Patients can continue receiving the same dose of irinotecan in the absence of major toxicity if before retreatment they fully recover from any non-hematological toxicity, absolute neutrophil count is 1500 microliters and platelet count is 100,000 microliters. Chemotherapy is discontinued on evidence of disease progression by RECIST version 1.1.

SECONDARY OUTCOMES:
Response rate | Every 2 cycles (every 8 weeks), from the beginning of the study until disease progression or death, which ever comes first (up to on average 60 months)
  Response rate is the number of patients with a partial response (by RECIST version 1.1) divided by the total number of patients.
Progression-free survival (PFS) | From beginning of the study until disease progression or death, which every comes first (up to on average 60 months)
  PFS is the time (in days) between study enrollment and disease progression (by RECIST version 1.1) or death, whichever comes first.
metastectomy (with curative intent) rate | Within 1 year of starting therapy
  Metastatectomy rate is the number of patients who undergo a surgical resection with curative intent divided by the total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sharma, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- Centro di Riferimento Oncologico, Aviano, Italy